CLINICAL TRIAL: NCT03240549
Title: Effectiveness and Safety of Adding Bevacizumab to Chemotherapy in Patients With Advanced Lung Adenocarcinoma With Stable Disease After 2 Cycles of First Line Combination Chemotherapy: a Multicenter, Prospective Cohort Study
Brief Title: Effectiveness and Safety of Adding Bevacizumab to First Line Chemotherapy in Lung Cancer Patients With Stable Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Bin Ai, Deputy chief physician, Beijing Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 121-2016007
Record Dates: First submitted 2017-07-20; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: advanced pulmonary adenocarcinoma; Bevacizumab; First line chemotherapy; Stable disease
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- conventional therapy group (No Intervention): Treatment with previous regimen of combined chemotherapy
- bevacizumab group (Experimental): Adding bevacizumab to the previous regimen of combined chemotherapy
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: bevacizumab — The patients in conventional group continued the previous chemotherapy,and the patients in experimental group received adding bevacizumab to previous chemotherapy regimen.
  Other Names: avastin
  Arms: bevacizumab group

SUMMARY:
Previous studies have shown that the addition of bevacizumab to the standard first-line platinum-based combination therapy can improve the objective response rate of patients with advanced non-squamous non-small cell lung cancer by 20% to 28% and improve survival. Data from these published literatures suggest that the improvement in objective response rates is due mainly to patients with stable disease of chemotherapy. It has been reported that 15% of patients achieved objective remission after continuing treatment with the regimen after receiving 2 cycles of platinum-based combination chemotherapy. Therefore, the use of 2 cycles of chemotherapy after stabilization of patients with bevacizumab, hoping to improve the objective response rate of such patients 20%, and may improve survival. For the above reasons, design this study to validate our hypothesis.

DETAILED DESCRIPTION:
Previous studies have shown that the addition of bevacizumab to the standard first-line platinum-based combination therapy can improve the objective response rate of patients with advanced non-squamous non-small cell lung cancer by 20% to 28% and improve survival. Data from these published literatures suggest that the improvement in objective response rates is due mainly to patients with stable disease of chemotherapy. It has been reported that 15% of patients achieved objective remission after continuing treatment with the regimen after receiving 2 cycles of platinum-based combination chemotherapy. Therefore, the use of 2 cycles of chemotherapy after stabilization of patients with bevacizumab, hoping to improve the objective response rate of such patients 20%, and may improve survival. For the above reasons, design this study to validate our hypothesis.

So a prospective cohort study has been designed to confirm this hypothesis, patients with advanced pulmonary adenocarcinoma who are stable after two cycles of platinum-based combination chemotherapy are objects of this study, and they can choose to continue the previous treatment regimen according to the guideline or adding bevacizumab to the regimen independently until the progression or intolerance of toxicity, or 4 to 6 cycles of chemotherapy in stable disease. The objective response rate in these two groups who received different treatment is the primary endpoint and the toxicity, quality of life, the progression free survival are the second endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. Age ≥18 years old, ≤75 years old;
3. Histologically or cytologically confirmed lung adenocarcinoma that can not treated with surgery with locally advanced (stage IIIb) or metastatic (IV) disease. Do not accept the diagnosis of lung adenocarcinoma alone based on sputum cytology;
4. Patients who have undergone targeted therapy for stage of disease (stage III, stage IV, stage IV) have not received treatment for advanced disease chemotherapy for patients with mutations associated with driving genes (eg, EGFR(epidermal growth factor receptor) mutations, ALK(anaplastic lymphoma kinase) gene fusion, etc.) could be included;
5. Patients who have received adjuvant or neoadjuvant therapy for non-metastatic lesions can be enrolled for more than 12 months at the beginning of the study treatment;
6. Patients who have measurable lesions according to RECIST 1.1;
7. First line chemotherapy is platinum combined with pemetrexed or paclitaxel;
8. Stable disease after 2 cycles chemotherapy;
9. Eastern Cooperative Oncology Group performance Status of 0 or 1;
10. Life expectancy ≥12 weeks;
11. There was no dose adjustment due to toxicity during the previous 2 cycles of combination chemotherapy;
12. The time delay is not more than 2 weeks due to toxicity of previous chemotherapy;
13. Adequate hematological function:ANC≥1.5 x 109/L，PLT≥100 x 109/L，Hb≥9 g/dL；
14. Adequate liver function:

    * Total bilirubin <1.5x ULN(the upper limit of the normal value), and
    * for patients without liver metastases, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 times ULN; for patients with liver metastases, both were less than 5 times ULN;
15. Adequate renal function:

    serum creatinine is equal to or less than 1.5 times ULN (upper limit of normal), - or creatinine clearance calculated value is greater than or equal to 60ml/min, and

    - routine urine urine protein negative or 24 hour urinary protein quantity is less than or equal to 1g;
16. Within 7 days before treatment, the international normalized ratio (INR) is less or equal to 1.5 times ULN, and partial thromboplastin time (PTT or aPTT) less than 1.5 times ULN;

Exclusion Criteria:

1. Mixed non-small cell and small cell carcinoma, large cell carcinoma, adenosquamous carcinoma;
2. Within 3 months before the election has a clear history of hemoptysis, that is, a single hemoptysis more than 2ml blood;
3. Images show signs of tumor invasion into the large blood vessels;
4. Patients with symptomatic central nervous system metastasis or intratumoral hemorrhage, the patient can not be selected regardless of whether or not to receive the relevant treatment;
5. Received chest radiotherapy within 28 days prior to enrollment;
6. Received a large number of surgical operations (including thoracotomy biopsy) or have a major trauma within 28 days prior to enrollment;
7. Current or resent (within the first 10 days of receiving the first dose bevacizumab) using aspirin (> 325 mg / day);
8. Current or recent (within the first 10 days of receiving the first dose bevacizumab) the use of full dose oral or parenteral anticoagulant or thrombolytic therapy.Allow prophylactic use of anticoagulants;
9. Medical history or examination results indicate that patients with hereditary bleeding tendency or coagulopathy may increase the risk of bleeding;
10. Uncontrolled hypertension (systolic blood pressure> 150 mmHg and / or diastolic blood pressure> 100 mmHg);
11. Previous hypertensive crisis or hypertensive encephalopathy patients;
12. Cardiovascular disease with clinical significance, including but not limited to CVA(cerebral vascular accident) or TIA（transient ischemic attack） (≤ 6 months before admission), myocardial infarction (≤ 6 months before enrollment), unstable angina, New York Heart Association classification ≥ Class II Congestive heart failure, need to be treated during the study and may interfere with the study of treatment, or drug can not control the serious arrhythmia;
13. Significant vascular disease (including but not limited to aortic aneurysm or proximal arterial thrombosis requiring surgery repair) within 6 months prior to enrollment;
14. Non-curative wounds, active peptic ulcers or fractures;
15. There was a history of abdominal fistula, gastrointestinal perforation, or intraperitoneal abscess within 6 months of enrollment;
16. Women who had a complete uterus (except for menopausal status over the last 24 months) during the six months after the study and at the last administration of bevacizumab, but did not use effective contraceptive methods (no contraindications to use background chemotherapy Drugs in the case of oral contraceptives, intrauterine devices, barrier contraceptives combined with spermicidal gels or sterilization surgery). During the study period and the last administration of bevacizumab within 90 days, men who did not agree to use effective contraceptive methods;
17. Pregnant and lactating women;
18. Received any other test medication or participated in another clinical trial within 28 days prior to enrollment;
19. Known hypersensitivity to bevacizumab or any of its excipients and any chemotherapeutic ingredients;
20. Signs of persistent or active infection requiring intravenous antibiotic therapy; other diseases, neurological or metabolic dysfunction; contraindications in the results of medical examination or laboratory findings or the use of a study drug or a patient at a high risk of treating the high risk associated with complications Suspicious disease or symptoms;
21. Tracheal - esophageal fistula or bronchial - pleural fistula;
22. Malignant tumor other than NSCLC within 5 years before enrollment, except for the adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer and ductal carcinoma in situ after radical resection;
23. Medical history or examination results showed thrombotic disease within 6 months before enrollment;
24. Patients with mental illness or no self-judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-08-31 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Assessment of the response should be done from the written consent to the 3 month after the last patient inrolled in the study, assessed up to 24 months.
  The percentage of patients who was assessed as complete response and partial response according RECIST (Response Evaluation In Solid Tumors).

SECONDARY OUTCOMES:
Duration of Response Duration of Response | The start point was the first remission until the date of first documented progression or date of death from any cause, which came first, assessed up to 30 months.
  The duration in responsive patients from the first remission to the progression.
Progression Free Survival. | The progression free survival was start from the written consent to the date of first documented progression or date of death from any cause, which came first,assessed up to 30 months.
  The time from the day written consent to the first date of objective progression or death from any cause.
Adverse Effects. | Assessment should be done from the written consent to the date 28 days after the last chemotherapy, assessed up to 24 months.
  The adverse effects of the treatment especially in hematology,cardiovascular system and renal system according the CTCAE 4.0, and the SAE(serious adverse events) in the treatment and follow up.
Quality of Life. | Assessment should be done from the written consent to the finish of this study, assessed up to 36 months.
  The quality of life should be assessed in the study using FACT-L(Functional Assessment of Cancer Therapy - Lung).

CONTACTS AND LOCATIONS:
Overall Officials: Yixin Zeng, Doctor, Study Chair — Beijing Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandler A, Gray R, Perry MC, Brahmer J, Schiller JH, Dowlati A, Lilenbaum R, Johnson DH. Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung cancer. N Engl J Med. 2006 Dec 14;355(24):2542-50. doi: 10.1056/NEJMoa061884. PMID 17167137
- [Derived] Ai B, Zhang L, Huang D, Chen J, Liu Z, Hu X, Zhou S, Hu Y, Zhao J, Yang F. Efficacy and safety of bevacizumab in advanced lung adenocarcinoma patients with stable disease after two cycles of first-line chemotherapy: A multicenter prospective cohort study. Thorac Cancer. 2020 Dec;11(12):3641-3644. doi: 10.1111/1759-7714.13687. Epub 2020 Oct 19. PMID 33073527